CLINICAL TRIAL: NCT04073264
Title: Isthmocele After Two Different Sutures in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 129/19
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Cesarean Scar Defect
MeSH Terms: interventions — Saran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monofilament (Experimental): monofilament absorbable suture
  Interventions: Procedure: monofilament
- polifilament (Active Comparator): synthetic absorbable braided (polifilament) suture
  Interventions: Procedure: monofilament

INTERVENTIONS:
Procedure: monofilament — In the intervention group,monofilament absorbable suture,will be used.

SUMMARY:
Cesarean delivery (CD) rates are rising globally. about 30% of women delivered by CD in 2015 only in the USA. This increasing CD rate has stimulated an interest in the potential short- and long-term morbidity of CD scars. In more than 50% of women with history of CD, a uterine scar defect, also called a "isthmocele," defined as a disruption of the myometrium in the CD uterine scar, can be observed when examined by gel instillation sonohysterography 6-12 months after the CD. Uterine scar defects detected on ultrasound have been associated with prolonged menstrual bleeding and postmenstrual spotting, as well as with an increased risk of several obstetrical complications in subsequent pregnancies, including uterine dehiscence and/or rupture, scar pregnancy and placenta previa and accreta. Another screening method associated with uterine scar rupture in women with prior CD is ultrasonographic measurement of the thickness of the lower uterine segment, as pioneered by Rozenberg et al. in 1996. A meta-analysis by Kok et al. supports the use of the residual myometrial thickness (RMT) for predicting uterine rupture during vaginal birth after cesarean. Uterine scar defects have been associated with lower RMT.

A growing body of evidence suggests that the surgical technique for uterine closure influences uterine scar healing and the RMT, but there is still no consensus about optimal uterine closure and type of suture. It is imperative to have evidence-based guidelines for each surgical step before recommending one technique over another.

The aim of our trial is to evaluate the incidence of cesarean scar defect according to type of suture at the time of cesarean

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton gestations
* Between ≥37 and ≤42 gestational age
* >18 <45 years
* Undergoing primary or secondary elective or urgent cesarean delivery

Exclusion Criteria:

* Multiple gestations
* Preterm cesarean
* 2 or more prior cesarean deliveries
* Uterine malformations
* Prior myomectomy
* Placenta accreta/previa

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 300 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
incidence of cesarean scar defects at ultrasound 6-months follow-up | 6-months follow-up after cesarean

SECONDARY OUTCOMES:
incidence of scar defects at hysteroscopy at 6 months follow-up | 6-months follow-up after cesarean
Symptoms of cesarean scar defect | 6-months follow-up after cesarean
  including pain, Abnormal bleeding, Vaginal discharge, Painful periods
RMT | 6-months follow-up after cesarean
  residual myometrial thickness at ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saccone G, De Angelis MC, Zizolfi B, Gragnano E, Musone M, Zullo F, Bifulco G, Di Spiezio Sardo A. Monofilament vs multifilament suture for uterine closure at the time of cesarean delivery: a randomized clinical trial. Am J Obstet Gynecol MFM. 2022 May;4(3):100592. doi: 10.1016/j.ajogmf.2022.100592. Epub 2022 Feb 4. PMID 35131497